CLINICAL TRIAL: NCT01491204
Title: Phase I Clinical Trial to Determine the Maximum Tolerated Dose and to Assess the Safety and Pharmacokinetic Profile of Oral Paclitaxel in Patients With Advanced Solid Cancer
Brief Title: Clinical Trial to Determine the Maximum Tolerated Dose and to Assess the Safety and Pharmacokinetic Profile of Oral Paclitaxel in Patients With Advanced Solid Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-OXL-101
Record Dates: First submitted 2011-12-05; First posted 2011-12-13 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- paclitaxel +HM30181 (Experimental)
  Interventions: Drug: Paclitaxel+HM30181

INTERVENTIONS:
Drug: Paclitaxel+HM30181 — oral, 3times for 4weeks

SUMMARY:
The main objective of this study is to determine the maximum tolerated dose (MTD) of Oral Paclitaxel. Eligible subjects of this study are patients with histologically or cytologically confirmed malignant solid tumor refractory to standard therapy.

Administration Schedule: 1 cycle of Oraxol®(paclitaxel+HM30181A) medication was 28 days and Oraxol® was administrated total 3 times once a week (day 1, 8, 15). The next cycle started on day 29.

Methods of Administration: HM30181A tablet was administered 1hour prior to the medication of paclitaxel

DETAILED DESCRIPTION:
Besides the main objective, there are 3 other objectives as follows.

To determine dose-limiting toxicity (DLT) Of Oraxol. To characterize the pharmacokinetics of HM30181A(pgp inhibitor), paclitaxel and its metabolites following oral administration of Oraxol.

To evaluate anticancer activity of Oraxol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must histologically or cytologically be diagnosed to have an advanced solid cancer.
2. Patients have progressive disease in spite of standard anti-cancer therapy or are not expected to benefit or prolong survival from any existing anti-cancer therapy
3. Patients who received chemotherapy, radiation therapy, surgery must have passed at least 4weeks since the final treatment and must have fully recovered from the toxicities Patients treated by Nitrosoureas or Mitomycin C must wait 6 weeks before becoming eligible.
4. ECOG performance status ≤ 2
5. Life expectancy ≥ 12 weeks
6. Patients have proper bone marrow, kidney, liver function and patients do not have remarkable dysfunction of heart and lung: WBC≥4000/mm3; Platelet ≥100,000/mm3; Hemoglobin≥9.0g/dL; ANC≥ 1,500 /mm3; Creatinine ≤ 1.5mg/dL; AST/ALT/ALP ≤ 3 X the upper limit of normal; Total bilirubin ≤2.0mg/dL *AST/ALT/ALP ≤ 3 X the upper limit of normal but <5 if liver or bone metastasis is present

Exclusion Criteria:

1. Patients with blood tumor (ex, leukemia), uncontrolled infectious disease, neurologic disorders, metastasis to CNS or ileus (patients requiring non-oral administration of anti-biotics to treat active bacterial infection are nor eligible, but patients can participate in the trial after complete eradication or control of the infection)
2. Patients who have received bone marrow transplant or are to receive bone marrow transplant.
3. Patients who had the medical history of atrial or ventricular arrhythmia or congestive heart failure or received medical treatment for myocardial infarction within 6 months.
4. Pregnant or lactating or with childbearing potential without use of adequate contraception (in case of men, appropriate contraception is required).
5. Patients who are on PGP inhibitor such as Cyclosporine or Verapamil which are prohibited.: Such patients may qualify after two-week wash-out period.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
MTD determination | Dose limiting Toxicity will be evaluated on Day 28 during Cycle 1